CLINICAL TRIAL: NCT04113473
Title: Effectiveness of Yoga Therapy for Neck Pain Relief in Patients With Cervical Spondylosis
Brief Title: An Evaluation of Yoga Therapy for Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Yog-Kulam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NMP/62548
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Cervical Spondylosis; Neck Pain
MeSH Terms: conditions — Spondylosis; Neck Pain | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): Experimental group received individualised yoga therapy twice a week for an hour for 12-weeks.
  Interventions: Other: Yoga Therapy
- Control Group (No Intervention): Control group were given education session and continued on usual care for 12-weeks.

INTERVENTIONS:
Other: Yoga Therapy — An hour of yoga therapy included loosening exercise (sukshma vyayama), yoga postures (asana), yoga breathing (pranayama), relaxation (shavasana) and meditation.
  Each participant were given handouts to follow home practice sessions everyday for twice a day for at least 15 minutes.
  Arms: Yoga Group

SUMMARY:
Cervical spondylosis is a chronic degenerative condition, commonly affecting >40-year-old adults worldwide. Cervical spondylosis is an important cause of neck pain and low back pain, and seriously affects the physical health, mental health, patients quality of life. Yoga has been most commonly used intervention for pain conditions. But its efficacy in cervical spondylosis has not yet been studied in clinical trials. The primary aim of the present study was to assess the efficacy of yoga chikitsa (therapy) compared with control intervention for neck pain caused by cervical spondylosis.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain of CS as per diagnostic criteria of International Classification of Diseases
* CS supported by a physical examination, and cervical radiographic examination
* History of neck pain longer than 3 months
* willing to provide informed consent

Exclusion Criteria:

* History of neck trauma, fracture or surgery,
* Systematic disease of the neck or spine including bones and joints conditions,
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Neck pain | Change from baseline to 12 weeks
  ain intensity was measured by a 10-cm VAS scale, with 0 = "no Pain" and 10 = "the worst imaginable pain

SECONDARY OUTCOMES:
Disability | Change from baseline to 12 weeks
  Neck disability was measured using neck disability index (NDI) score
Health related Quality of Life | change from baseline to 12 weeks
  Short Form-36 assessed the Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Yog-Kulam; Shekhar Sharma, Study Director — NMP Medical Research Institute, India; Jaydeep Joshi, Study Chair — Yog-Kulam
Locations (1):
- Pain Clinic, NMP Medical Research Institute, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided